CLINICAL TRIAL: NCT05850000
Title: Dementia Clinical Trials: A Study on the Clinical Trial Participation of Dementia Patients
Brief Title: Discovering Factors in the Clinical Trial Journey of Dementia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 94341447
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Dementia
Keywords: dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to collect comprehensive data on the clinical trial experience of dementia patients. Its goal is to identify the factors that limit patients' ability to join or complete a trial successfully. Clinical trial participation often favors specific demographic groups, and limited research exists on the impact of trial attributes on participation. Therefore, this study aims to analyze data from various demographic groups and identify any recurring trends that could provide valuable insights for future dementia patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Participant has a diagnosis of dementia.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Enrolled in another research study
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dementia who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a dementia clinical study. | 3 months
Number of dementia patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perng CH, Chang YC, Tzang RF. The treatment of cognitive dysfunction in dementia: a multiple treatments meta-analysis. Psychopharmacology (Berl). 2018 May;235(5):1571-1580. doi: 10.1007/s00213-018-4867-y. Epub 2018 Mar 3. PMID 29502274
- [Background] Whitehouse PJ, Kittner B, Roessner M, Rossor M, Sano M, Thal L, Winblad B. Clinical trial designs for demonstrating disease-course-altering effects in dementia. Alzheimer Dis Assoc Disord. 1998 Dec;12(4):281-94. doi: 10.1097/00002093-199812000-00007. PMID 9876956
- [Background] Graham NS, Sharp DJ. Understanding neurodegeneration after traumatic brain injury: from mechanisms to clinical trials in dementia. J Neurol Neurosurg Psychiatry. 2019 Nov;90(11):1221-1233. doi: 10.1136/jnnp-2017-317557. Epub 2019 Sep 21. PMID 31542723

DOCUMENTS (1):
  • Informed Consent Form (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT05850000/ICF_000.pdf